CLINICAL TRIAL: NCT02203318
Title: Can the Hypertrophy of Contralateral Testis Predict the Absence of the Non-palpable Testis in the Boys Aged From 6months to 18months of Age ?
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2014-0385
Record Dates: First submitted 2014-07-27; First posted 2014-07-29 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Focus of Study
Keywords: cryptorchidism, undescended testis, hypertrophy of contralateral testis
MeSH Terms: conditions — Cryptorchidism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- control: healthy children with normal bilateral testis
- undescended palpable testis: patient whose affected testis is not descended to the normal position but palpable and exist intact in the upper area
- non-paplpable testis: patient whose affected testis is not palpable during the physical examination

SUMMARY:
The aim of this study is to verify whether the hypertrophy of contralateral testis may predict the absence of the non-palpable testis in the boys younger than 24months of age. According to the previous studies of other countries, the large size of the contralateral testis of the nonpalpable testis has positive correlation woth the weak viability of the affected testis. We are going to evaluate this hypothesis with prospective study. 3 groups are going to be enrolled into this study ; non-palpable testis group(Group1), palpable but not normally descended testis group(group2) and control group(group3). The size of testis will be measured with Ultrasound and the length, width and the height will be measured before surgery at outpatient department. For the group 1 & 2, the viability of the affected testis will be evaluated and compared after surgery. In addition the comparison with normal control group is also going th be conducted.

ELIGIBILITY:
Inclusion Criteria:

1. neonates or Infants who visited the out-patient clinic with nonpalpable or undescended testis.(group 1, 2) aged from 6months to 18months
2. neonates or Infants aged from 6months to 18months with normal testis (volunteers, Group3)

Exclusion Criteria:

1. previous history of hormonal therapy.
2. chromosomal abnormality
3. previous history of abdomen or inguinal area surgery
4. children diagnosed with epididymitis or orchitis
5. twin baby
6. infants with premature (<37 weeks) birth history

Ages: 6 Months to 18 Months | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Study Population: totally, 72 children : unpalpable testis : 24 children, palpable undescended testis : 24 children, normal control : 24 children
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2014-07; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Size of contralateral testis | 1 day of initial visit
  The testicular size is measured 3-dimensionally with ultrasonography. The length, width and height will be measured and the volume of testis will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Yonsei University College of Medicine, Seoul, Seoul, South Korea